CLINICAL TRIAL: NCT05851716
Title: A Prospective, Single-arm, Single-center Observational Study to Evaluate the Clinical Effectiveness of an Intelligent Reporting System for the Upper Gastrointestinal Endoscopy
Brief Title: Upper Gastrointestinal Endoscopy Reporting System in Improving Report Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: EA-23-006
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Endoscopy, Gastrointestinal; Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of an AI-based reporting system for upper gastrointestinal endoscopy. The main question it aims to answer is: Whether the AI-based reporting system can improve the completeness of the reports, which are drafted by endoscopists with the AI assistance. Participants will undergo upper gastrointestinal endoscopy examination as routine. The junior endoscopists will draft the report with the assiatance of the AI system. And the senior and expert endoscopists will draft the report using the traditional reporting system without AI assistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years
2. Aim to undergo screening, surveillance, and diagnosis
3. Undergo sedated EGD
4. Able to read, understand, and sign informed consent

Exclusion Criteria:

1. EGD contraindications
2. Not suitable for sedated endoscopy after anaesthesia evaluation
3. Biopsy contraindications
4. Active upper gastrointestinal bleeding or emergency oesophagogastroduodenoscopy (EGD)
5. Pregnancy
6. Upper gastrointestinal surgery or residual stomach
7. Not suitable for recruitment after investigator evaluation because of other high-risk conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is not limited. Patients aim to undergo screening, surveillance, and diagnosis upper gastrointestinal endoscopy will be accessed for eligibility.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Completeness of reporting lesions | one month
  Calculation method = number of report lesions / total number of lesions x 100%

SECONDARY OUTCOMES:
Completeness of report drafting on lesion features | one month
  Calculation method = number of drafted features of lesions / total number of features required to be drafted x 100%
Accuracy of report drafting on lesion features | one month
  Calculation method = number of accurately drafted features of lesions / total number of drafted features x 100%
Reporting time | one month
  The time that endoscopists draft reports
Completeness of reporting lesions of AI system | one month
  Calculation method = number of report lesions / total number of lesions x 100%
Accuracy of report drafting on lesion features of AI system | one month
  Calculation method = number of accurately drafted features of lesions / total number of drafted features x 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No